CLINICAL TRIAL: NCT06616246
Title: Evaluating the Use of Community Members Trained as Health Coaches to Deliver the HealthyLifetimeTM Program
Brief Title: Training Community Members to be Coaches to Deliver the HealthyLifetime Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Potempa, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-PAF04327
Record Dates: First submitted 2024-09-12; First posted 2024-09-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Health Behaviors; Functional Decline; Chronic Disease; Risk Factors
Keywords: health coach; health resiliency; independent self-care; community health workers; independent aging
MeSH Terms: conditions — Health Behavior; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Coach (Active Comparator): HealthyLifetime program is administered by an experienced nurse coach.
  Interventions: Behavioral: HealthyLifetime
- Health worker coach (Experimental): HealthyLifetime program is administered by a community health worker
  Interventions: Behavioral: HealthyLifetime

INTERVENTIONS:
Behavioral: HealthyLifetime — HealthyLifetimeTM [HL] seeks to intervene early in the aging process when individuals have the best chance for longer-term benefits of changing their health behavior, staving off functional decline, and minimizing the onset or exacerbation of chronic conditions.

SUMMARY:
The goal of this randomized controlled study is to learn if, in addition to nurses, community members can be trained as health coaches to deliver the HealthyLifetime (HL) program to people without complex chronic health conditions, an intervention that provides a short-term and effective health coaching intervention delivered through a virtual platform to improve health, resiliency, and independent self-care to participants who are without complex chronic conditions. The main question it aims to answer is:

• Can Community Health Coaches achieve the same level of competency and outcome as Nurse Health Coaches in participants without complex chronic conditions?

DETAILED DESCRIPTION:
The investigators will evaluate the use of trained community members [Health Coach, (HC)] in delivering the HealthyLifetime program to adults without complex chronic conditions. Our cumulative learnings about effective HL strategies, training, and outcomes assessments set the stage for the proposed use of trained community members as HL Health Coaches under the supervision of the nurse Clinical Services Manager. The Independent Living Index (ILI) measures 'risk' for loss of independence due to functional decline from complex chronic conditions and other factors. The investigators will use the ILI and other medical information to determine which participants can be appropriately delegated to non-clinical staff coaches, which the investigators define as participants without complex chronic conditions. Our training methods will be adapted for use with community members. Our health coaching competency assessment tools will be used to measure community members trained as Health Coaches and Nurse Health Coach' relative competency. The investigators will compare quantitative and qualitative outcomes between participants coached by HL Health Coaches (community members) vs. HL Nurse Health Coaches and any outcome differences due to demographic, social determinants, or other factors. Finally, the investigators intend to evaluate the program satisfaction and potential cost impact using our Medical Use Index as a proxy for cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 30 years of age, with no more than three, uncomplicated chronic conditions and want to learn to take better care of their health.
* Independent Living Index (ILI) greater than 35. ILI is derived by averaging the outcome measures scores.
* A score of less than 4 on items related to anxiety and depressive symptoms
* Have Medicare and/or Medicaid insurance.
* Be able to read, speak, and hear English - but may use glasses or hearing aids, if needed;
* Tell us their age, date of birth, address, and phone number, and explain their health problems;
* Have a computer, iPad (Tablet), or Smartphone with an Internet connection, email address, a working camera, and microphone;
* Be able to use their computer/tablet to connect to video chat sessions like Zoom in a private space in their home or a private room
* Are not currently participating in any other studies involving diet, weight management, exercise and/or coaching at the current time; and
* Reside in Michigan.

Exclusion Criteria:

* ● Are less than 30 years of age.

  * Have more than three, uncomplicated chronic conditions.
  * A score of more than 4 on items related to anxiety and depressive symptoms
  * Do not have Medicare and/or Medicaid insurance.
  * Do not reside in Michigan.
  * Have a new acute health problem that requires seeing a doctor more than once a month for acute medical treatment.
  * Have been told their illness is not curable.
  * Need help remembering their name, date of birth, or health problems.
  * Cannot use glasses or a hearing aid to see or hear well enough to read materials on the computer or talk to the nurse easily.
  * Are currently participating in any other studies involving diet, weight management, exercise and/or coaching at the current time; and
  * Do not have, or cannot use, a computer, iPad, or another device with the Internet at home to use Zoom (e.g., internet streaming).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Participant Self- rated satisfaction with various aspects of their home and neighborhood. | At 0, 8 and 20 weeks after study enrollment.
  Participants perception of their home and neighborhood on a scale of 1= Extremely Satisfied to 5 = Not at all satisfied
Satisfaction with Quality of Life | At 0, 8 and 20 weeks after study enrollment.
  Questions are about how participant experiences their quality of life on a scale where "1" = "Do not agree at all" and "5" = "Agree completely",
Positive and negative Lifestyle Habits aggregate | At 0, 8 and 20 weeks after study enrollment.
  Composite score of activities that participants engage in that affect health in a negative (lower score) or positive way (higher score) on a scale of 1 to 5. Smoking (yes or no), alcohol (number of drinks per week, 5= none, 5= more than eight), exercise (1 = none to 5= more than 3 hours/week), food choices (One serving or less a day to 5 or more servings a day of positive, e.g., vegetable, or negative food choice, e.g., sugary food), amount of sleep (1 = less than 4 to 5 = more than 7 hours)
Change in Goal attainment score | At 0, 8 and 12 weeks after study enrollment.
  Health goals of participants (up to 3) confidence in achieving goal (1= Not confident at all to 10 = Completely Confident)
Change in Self-efficacy in ability to continue essential life activities | At 0, 8 and 20 weeks after study enrollment.
  Ability or confidence of the participant in doing certain activities on a scale of 1= Cannot do this myself/Not confident at all to 5 = Always able to do myself/Completely Confident. For the purposes of answering these questions, confidence is defined as the belief in the participant's chances of being able to do and/or complete an activity (e.g., hobbies and recreation, social visits, chores, errands, etc.) or task (e.g., hobbies and recreation, social visits, chores, errands, etc.) successfully however the participant defines it.

SECONDARY OUTCOMES:
Change in Sustained higher values of primary measures at 3 months | 20 weeks after study enrollment
  Are effects of program noted at 8 weeks still present at 20 weeks.
Change in Self-reported medical visits | At 0, 8 and 20 weeks after study enrollment.
  Number of unplanned medical visits with doctor or primary medical provider in past 2 months (0 to 10), emergency room visits (0 to 10 ), overnight stay in hospital (0 to 10).

OTHER OUTCOMES:
CONFIDENCE IN MANAGING SYMPTOMS | At 0, 8 and 20 weeks after study enrollment.
  Participant indicate confidence or certainty NOW that they can do the activity or task on scale scale where "1" = "Not confident" and "5" = "Very confident,"
PHYSICAL SYMPTOM INVENTORY | At 0, 8 and 20 weeks after study enrollment.
  Participant indicates how often they experienced physical symptoms IN THE LAST WEEK on a scale where "1" = "Rarely" and "5" = "Almost always"

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Potempa, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No